CLINICAL TRIAL: NCT02409472
Title: A Randomized Trial Of Intensive Versus Minimal Surveillance Of Patients With Resected Dukes B2-C Colorectal Carcinoma
Brief Title: Intensive Versus Minimal Surveillance of Patients With Resected Dukes B2-C Colorectal Carcinoma
Acronym: GILDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GILDA
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer; Surveillance
Keywords: randomized clinical trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- minimal surveillance (Other): Minimal program for colon cancer: Office visit and CEA at 4,8,12,16,20,24,30,36,42,48, and 60 months. Colonoscopy at 12, and 48 months. Liver echography* at 8, and 20 months.
  Interventions: Other: surveillance program after completion of primary treatment
- intensive surveillance (Other): Intensive program for colon cancer: Office visit, complet blood count (CBC), CEA+ Carbohydrate Antigen (CA) 19.9 at 4,8,12,16,20,24,30,36,42,48, and 60 months. Colonoscopy at 12, 24, 36, 48,and 60 months. Liver echography* at 4,8,12,16,24,36,48, and 60 months. Chest X-ray at 12,24,36,48,and 60 months.
  Interventions: Other: surveillance program after completion of primary treatment

INTERVENTIONS:
Other: surveillance program after completion of primary treatment — These are two different surveillance programs for Dukes B2-C colorectal cancer patients who have no evidence of disease at the end of their front line treatment (surgery and adjuvant radio-chemotherapy, if indicated). These programs differ greatly in the frequency of diagnostic imaging. They had similar schedules of physical examinations and carcinoembryonic antigen (CEA) assessments.

SUMMARY:
Dukes B2-C colorectal cancer patients who had no evidence of disease at the end of their front line treatment (surgery and adjuvant radio-chemotherapy, if indicated) are eligible for the trial and randomized to two different surveillance programs. These programs differ greatly in the frequency of diagnostic imaging. They have similar schedules of physical examinations and carcinoembryonic antigen (CEA) assessments. Patients will receive baseline and yearly health-related quality of life (HR-QoL) questionnaires. Primary outcomes are overall survival and QoL.

DETAILED DESCRIPTION:
Minimal program for colon cancer: Office visit and CEA at 4,8,12,16,20,24,30,36,42,48, and 60 months. Colonoscopy at 12, and 48 months. Liver echography* at 8, and 20 months.

Intensive program for colon cancer: Office visit, CBC, CEA+CA 19.9 at 4,8,12,16,20,24,30,36,42,48, and 60 months. Colonoscopy at 12, 24, 36, 48,and 60 months. Liver echography* at 4,8,12,16,24,36,48, and 60 months. Chest X-ray at 12,24,36,48,and 60 months.

* Abdominal-pelvis C.T., as an alternative to echography, was a 2° level exam only (doubtful results of physical examination or echography; increasing levels of CEA; predictable poor sensitivity of echography due to obesity or other anatomic-clinical conditions)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven adenocarcinoma of the colon or rectum with Dukes Astler-Coller modification stage B2-C who had been treated with curative intent (radical excision ± adjuvant radio-chemotherapy) .
* Eligible patients had to be free of known cancer prior to study entry as attested by negative results of endoscopy, liver ultrasonography, chest roentgenography and serum CEA level performed < 4 months before randomization

Exclusion Criteria:

* Inability to undergo testing (disability, allergy to contrast agents, etc.) and patients geographically not amenable to full follow-up.
* Patients enrolled onto any other research protocol that requires strict adherence to any specific follow-up practice.
* A history of any previous malignancy in the last 10 years (other than carcinoma in situ of the cervix or non-melanoma skin cancer).
* No informed consent to participate in the trial according to local regulatory guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 1998-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5-year OS
  OS is defined as the time from randomization to death from any cause
Health Related Quality of Life | Yearly assessment over 5 years
  mean scores for Short Form Health Status Survey (SF)12 and Psychological General Well-Being (PGWB) questionnaires

SECONDARY OUTCOMES:
Disease free survival (DFS) | 5-year DFS
  DFS is defined as the time from randomization to the earliest occurrence of progression or second primary colorectal cancer in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Andreoni, MD, Study Chair — European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Rosati G, Ambrosini G, Barni S, Andreoni B, Corradini G, Luchena G, Daniele B, Gaion F, Oliverio G, Duro M, Martignoni G, Pinna N, Sozzi P, Pancera G, Solina G, Pavia G, Pignata S, Johnson F, Labianca R, Apolone G, Zaniboni A, Monteforte M, Negri E, Torri V, Mosconi P, Fossati R; GILDA working group. A randomized trial of intensive versus minimal surveillance of patients with resected Dukes B2-C colorectal carcinoma. Ann Oncol. 2016 Feb;27(2):274-80. doi: 10.1093/annonc/mdv541. Epub 2015 Nov 16. PMID 26578734